CLINICAL TRIAL: NCT06934603
Title: Microplastic Exposure From Clear Aligner Wear: An In Vivo, Longitudinal Study of Orthodontic Patients
Brief Title: Microplastic Exposure From Clear Aligner Wear (MPE)
Acronym: MPE
Status: Recruiting | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 25-0426
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Microplastic Exposure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study will collect and retain saliva and urine samples at each of 3 time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Clear Aligner Treatment: Orthodontic patients already scheduled to receive clear aligner treatment at UNC Orthodontic clinics.
  Interventions: Other: Clear Aligner Treatment

INTERVENTIONS:
Other: Clear Aligner Treatment — This study is observational. Only patients who are previously scheduled to receive clear aligner treatment from their orthodontic provider will be recruited.

SUMMARY:
An observational longitudinal study measuring microplastic exposure and physiologic uptake in orthodontic patients receiving clear aligner treatment.

DETAILED DESCRIPTION:
This study is investigating whether orthodontic patients already scheduled to receive clear aligner treatment have changes in their microplastic exposure and physiologic uptake pre- and post-treatment. Consented and enrolled participants will provide unstimulated saliva and urine samples at three timepoints before regularly scheduled orthodontic appointments: Pre-treatment (Visit 1), 6-12 weeks post-treatment (Visit 2), and 16-24 weeks post-treatment (Visit 3). The saliva and urine samples will be filtered and then analyzed for microplastic content using mass spectroscopy, Raman spectroscopy and scanning electron microscopy approaches.

ELIGIBILITY:
Inclusion Criteria:

* Individuals (all sexes, genders, races, and ethnicities) aged at least 10 years (in adult dentition) and at most 75 years
* Receiving comprehensive, Phase II orthodontic treatment with clear aligner therapy
* Stable physical health (ASA I or II), as determined by study coordinator or PI
* Able to comprehend and follow requirements of study (including availability on scheduled visit dates)
* Patient and parental consent (and assent for minors) for participation in the study

Exclusion Criteria:

* Receiving orthodontic treatment with fixed appliances
* Receiving hybrid treatment with fixed appliances and aligners
* Receiving Phase I orthodontic treatment with fixed appliances
* Established history of severe xerostomia (dry mouth), severe periodontal disease with actively bleeding gums, significant oral abrasions/ulcers or growths, current alcohol abuse, and/or recreational drug abuse
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase risk associated with participation
* Drinking, eating, or brushing teeth within 1 hour of study visit
* Removing aligners within 1 hour of study visit
* Developmental or cognitive disability such that the patient cannot self-consent, comprehend, and follow the requirements of the study based on research site personnel's assessment

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes patients identified from UNC orthodontic clinics who are scheduled (prior to study engagement) to receive clear aligner treatment.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2035-07-01 (Estimated); Study Completion 2035-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in salivary microplastic abundance over time. | Pre-treatment through 16-24 weeks post-treatment.
  Differences in microplastic abundance in saliva collected pre-treatment with clear aligners, 6-12 weeks post-treatment, and 16-24 weeks post-treatment.
Change in urinary microplastic abundance over time. | Pre-treatment through 16-24 weeks post-treatment.
  Differences in microplastic abundance in urine collected pre-treatment with clear aligners, 6-12 weeks post-treatment, and 16-24 weeks post-treatment.

SECONDARY OUTCOMES:
Change in salivary microplastic size over time. | Pre-treatment through 16-24 weeks post-treatment.
  Differences in microplastic size in saliva collected pre-treatment with clear aligners, 6-12 weeks post-treatment, and 16-24 weeks post-treatment.
Change in salivary microplastic composition over time. | Pre-treatment through 16-24 weeks post-treatment.
  Differences in microplastic identities in saliva collected pre-treatment with clear aligners, 6-12 weeks post-treatment, and 16-24 weeks post-treatment.
Change in urinary microplastic size over time. | Pre-treatment through 16-24 weeks post-treatment.
  Differences in microplastic size in urine collected pre-treatment with clear aligners, 6-12 weeks post-treatment, and 16-24 weeks post-treatment.
Change in urinary microplastic composition over time. | Pre-treatment through 16-24 weeks post-treatment.
  Differences in microplastic identities in urine collected pre-treatment with clear aligners, 6-12 weeks post-treatment, and 16-24 weeks post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Jacox, DMD, PhD, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: Beginning 9 and continuing for 36 months following publication.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC